CLINICAL TRIAL: NCT04273906
Title: End-range Mobilization Effecting Pressure Pain Threshold in Knee Osteoarthritis
Brief Title: End-range Mobilization on Pressure Pain Threshold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MaitlandKneePPT
Record Dates: First submitted 2020-02-12; First posted 2020-02-18 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Knee Osteoarthritis
Keywords: Musculoskeletal Manipulations; Osteoarthritis, Knee; Pain Threshold
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- End-range mobilization (Experimental): End-range mobilization performed in end-position of the tibiofemoral joints' flexion and extension for 2*3 min
  Interventions: Procedure: End-range mobilization; Procedure: Placebo technique
- Placebo (Placebo Comparator): Hands-on treatment technique performed in end-range of the tibiofemoral joints' flexion and extension for 2*3 min
  Interventions: Procedure: End-range mobilization; Procedure: Placebo technique

INTERVENTIONS:
Procedure: End-range mobilization — End-range mobilization performed in end-range of the tibiofemoral joints' flexion and extension
Procedure: Placebo technique — Hands-on technique performed in end-range of the tibiofemoral joints' flexion and extension

SUMMARY:
Pain in knee osteoarthritis (OA) represents increased pain intensity due to peripheral and central sensitivity. Pressure pain threshold (PPT) is a widely applied (used) method for measuring the magnitude of peripheral and central sensitivity in knee OA. Among several manual therapy techniques increasing PPT in knee OA, the effect of end-range mobilization has not been evaluated so far. The aim of this study was to investigate the immediate effect of end-range mobilization compared to placebo on increase of PPT and some function-related measures.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is the most common form of arthritis contributing to a major cause of disability worldwide. Although many mechanisms may contribute to knee pain severity, the patient-reported hyperalgesia can be attributed to peripheral and central sensitivity in knee OA. Pressure pain threshold (PPT) measurement is a simple and commonly applied method for measuring somatosensory function in musculoskeletal disorders, just as in knee OA. Many trials have shown a lower PPT value in knee OA underlining the presence of peripheral and central sensitivity compared to healthy controls.

Manual therapy techniques, as a preferred treatment option, may not only alleviate pain, but also increase pain tolerance to locally applied mechanical pressure. Positive results of different manual therapy techniques on increase of PPT has been reported in knee OA. End-range manual therapy is an option for the decrease of sensitivity in knee OA; however, the effect of end-range mobilization has not been evaluated so far in knee OA.

ELIGIBILITY:
Inclusion Criteria:

* the clinical classification criteria of knee OA according to the American College of Rheumatology
* Categorization of patients as End Of Range Problem based on Maitland manual therapy
* female patients aged between 60 and 80 years
* uni/bilateral moderate-to-severe symptomatic tibiofemoral knee osteoarthritis with radiographic evidence of Kellgren-Lawrence scale 2 or 3
* pain during weight-bearing activities at least within 6 months
* at least 90° knee flexion
* sufficient mental status.

Exclusion Criteria:

* acute inflammation of the knee
* total knee replacement in the opposite side
* severe degenerative lumbar spine disease (e.g. spondylolisthesis)
* systemic inflammatory arthritic or neurological condition
* physiotherapy/balneotherapy attendance or manual therapy within 3 months
* intraarticular injections in the prior 12 months
* use of walking aids
* contraindication for manual therapy
* complex regional pain syndrome
* cognitive impairment

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients are enrolled due to patient characteristics from other study
Enrollment: 40 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
PPT of the knee | 30 minutes
  pressure pain threshold at the knee

SECONDARY OUTCOMES:
PPT of the m. Extensor Carpi Radialis Longus (ECRL) | 30 minutes
  pressure pain threshold at the ECRL
General Pain Intensity | 30 minutes
  General Pain Intensity measured with Visual Analogue Scale (VAS)
Timed Up and Go test | 30 minutes
  Timed Up and Go test measuring functional capacity
Pain intensity during Timed Up and Go test | 30 minutes
  associated pain intensity during the Timed Up and Go test
Passive tension of the knee | 30 minutes
  Passive tension of the knee at the beginning of pain

CONTACTS AND LOCATIONS:
Overall Officials: Miklós Pozsgai, Study Chair — Zsigmondy Vilmos Spa and Balneological Hospital of Harkány
Locations (1):
- Miklós Pozsgai, Harkány, Please Select, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kidd BL. Osteoarthritis and joint pain. Pain. 2006 Jul;123(1-2):6-9. doi: 10.1016/j.pain.2006.04.009. Epub 2006 May 22. No abstract available. PMID 16714085
- [Background] Wise BL, Niu J, Zhang Y, Wang N, Jordan JM, Choy E, Hunter DJ. Psychological factors and their relation to osteoarthritis pain. Osteoarthritis Cartilage. 2010 Jul;18(7):883-7. doi: 10.1016/j.joca.2009.11.016. Epub 2010 Mar 24. PMID 20346403
- [Background] Bajaj P, Bajaj P, Graven-Nielsen T, Arendt-Nielsen L. Osteoarthritis and its association with muscle hyperalgesia: an experimental controlled study. Pain. 2001 Aug;93(2):107-114. doi: 10.1016/S0304-3959(01)00300-1. PMID 11427321
- [Background] Imamura M, Imamura ST, Kaziyama HH, Targino RA, Hsing WT, de Souza LP, Cutait MM, Fregni F, Camanho GL. Impact of nervous system hyperalgesia on pain, disability, and quality of life in patients with knee osteoarthritis: a controlled analysis. Arthritis Rheum. 2008 Oct 15;59(10):1424-31. doi: 10.1002/art.24120. PMID 18821657
- [Background] Wylde V, Palmer S, Learmonth ID, Dieppe P. Somatosensory abnormalities in knee OA. Rheumatology (Oxford). 2012 Mar;51(3):535-43. doi: 10.1093/rheumatology/ker343. Epub 2011 Nov 24. PMID 22120461
- [Background] Hendiani JA, Westlund KN, Lawand N, Goel N, Lisse J, McNearney T. Mechanical sensation and pain thresholds in patients with chronic arthropathies. J Pain. 2003 May;4(4):203-11. doi: 10.1016/s1526-5900(03)00557-1. PMID 14622705
- [Background] Kaya Mutlu E, Ercin E, Razak Ozdincler A, Ones N. A comparison of two manual physical therapy approaches and electrotherapy modalities for patients with knee osteoarthritis: A randomized three arm clinical trial. Physiother Theory Pract. 2018 Aug;34(8):600-612. doi: 10.1080/09593985.2018.1423591. Epub 2018 Jan 8. PMID 29308949
- [Background] Khademi-Kalantari K, Mahmoodi Aghdam S, Akbarzadeh Baghban A, Rezayi M, Rahimi A, Naimee S. Effects of non-surgical joint distraction in the treatment of severe knee osteoarthritis. J Bodyw Mov Ther. 2014 Oct;18(4):533-9. doi: 10.1016/j.jbmt.2013.12.001. Epub 2013 Dec 11. PMID 25440203